CLINICAL TRIAL: NCT04949633
Title: Oxytocine Versus Prostaglandines Pour le déclenchement du Travail Des Femmes Dont le Col Est défavorable après 24 Heures de Maturation Cervicale : Essai Multicentrique randomisé de Non infériorité
Brief Title: Oxytocin vs Prostaglandins for Labor Induction of Women With an Unfavorable Cervix After 24h of Cervical Ripening
Acronym: OPIC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DR200090; 2021-000989-15 (EudraCT Number)
Record Dates: First submitted 2021-06-03; First posted 2021-07-02 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cervical Ripening; Unfavorable Cervix
Keywords: cervical ripening; oxytocin; prostaglandin; cesarean delivery
MeSH Terms: interventions — Prostaglandins; Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction of labor (Experimental): women randomized in the experimental group will be admitted to the labor ward to undergo induction of labor with intra-veinous oxytocin and early amniotomy. Oxytocin will be administered according to the French guidelines for induction of labor. Maximum oxytocin used should not exceed 10 UI.
  Interventions: Drug: Oxytocin
- Second cervical ripening (Active Comparator): women randomized in the control group will undergo a second cervical ripening lasting a maximum of 24 hours with either:
  * Vaginal slow releasing system of dinoprostone PROPESS® which is inserted in the vagina, against the cervix and left in place during 24 hours.
  * Oral misoprostol (ANGUSTA®) 25 µg every 2 hours, 8 times (maximum dosage should not exceed 200µg). Tablets will be given one at the time by midwives.
  * Vaginal gel of dinoprostone (2 mg PROSTINE®) every 6 hours, maximum dose of 6 mg.
  The choice of the cervical ripening agent will depend of the local protocol of the participating maternity unit. The choice between ANGUSTA®, PROPESS® and PROSTINE® will be made by investigators of each participating unit at the beginning of the trial.
  At the end of the second cervical ripening procedure women not in labor will be transferred to the labor ward for induction of labor with oxytocin.
  Interventions: Drug: Prostaglandins; Drug: Oxytocin

INTERVENTIONS:
Drug: Prostaglandins — Second cervical ripening lasting a maximum of 24 hours
  Arms: Second cervical ripening
Drug: Oxytocin — Induction of labor with oxytocin.

SUMMARY:
Twenty-two percent of deliveries in France are induced. In cases where labor is induced and cervix is unfavorable, cervical ripening prior oxytocin administration is advised in order to reduce the risk of cesarean delivery. Cervical ripening agents, pharmacological (prostaglandins) or mechanical are administered during 24 hours. After 24 hours, most women will be either delivered or in labor but 25% of women will require further induction of labor. For 16% of women who undergo cervical ripening, whatever the cervical ripening method, the cervix remains unchanged after 24 hours. The management of these women is not consensual and depends on the maternity unit where women are cared for.

This study seeks to identify the most appropriate strategy for the management of women with an unfavorable cervix after 24 hours of cervical ripening, a strategy which would be associated with the lowest maternal and perinatal morbidity but also with the best maternal satisfaction. Because both strategies are practiced in France, the trial would compare: induction of labor with oxytocin and repeated cervical ripening. The aim is to show that repeating cervical ripening is an unnecessary procedure. And more specifically that oxytocin administration is not associated with a higher caesarean delivery rate and that it reduces the time to delivery in comparison with cervical ripening with prostaglandins.

DETAILED DESCRIPTION:
Twenty-two percent of deliveries in France are induced. In cases where labor is induced and cervix is unfavorable, cervical ripening prior oxytocin administration is advised in order to reduce the risk of cesarean delivery. Cervical ripening agents, pharmacological (prostaglandins) or mechanical are administered during 24 hours. After 24 hours, most women will be either delivered or in labor but 25% of women will require further induction of labor. For 16% of women who undergo cervical ripening, whatever the cervical ripening method, the cervix remains unchanged after 24 hours. The management of these women is not consensual and depends on the maternity unit where women are cared for. In some units, women are admitted into labor ward for induction of labor with oxytocin. Elsewhere cervical ripening is repeated in order to obtain a favorable cervix and to reduce the risk of caesarean delivery.

This study seeks to identify the most appropriate strategy for the management of women with an unfavorable cervix after 24 hours of cervical ripening, a strategy which would be associated with the lowest maternal and perinatal morbidity but also with the best maternal satisfaction. Because both strategies are practiced in France, the trial would compare: induction of labor with oxytocin and repeated cervical ripening. The policy of induction of labor with oxytocin, being the simpler strategy, would be acceptable if it did not lead to a substantially proportion of women with caesarean deliveries compared with a second cervical ripening. This multicenter non inferiority randomized trial will recruit women with an unfavorable cervix (bishop score ≤ 6) after 24 hours of cervical ripening (pharmacological or mechanical) and randomize them to either induction of labor with oxytocin or to a second cervical ripening with prostaglandins. The aim is to show that repeating cervical ripening is an unnecessary procedure. And more specifically that oxytocin administration is not associated with a higher caesarean delivery rate and that it reduces the time to delivery in comparison with cervical ripening with prostaglandins.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* ≥ 18 years old
* With a singleton cephalic pregnancy
* ≥37+0 weeks of gestation
* Gestational age estimated from the first trimester ultrasound (realized between 11+0 and 13+6 weeks of gestation)
* With a medical indication of labor with a previous pharmacological or mechanical cervical ripening of 24 hours
* Bishop score ≤ 6 at inclusion (unfavorable cervix)
* French health insurance policy holder
* Written informed consent

Exclusion Criteria:

* Any measures of legal protection
* Prior caesarean section or uterine scar
* Contra-indications to a vaginal delivery
* Foetus with suspected severe congenital abnormalities
* Pathological foetal heart rate
* Contra-indications to ANGUSTA® (oral misoprostol, cervical ripening agent)
* Contra-indications to PROPESS® (vaginal slow releasing system of dinoprostone, cervical ripening agent)
* Contra-indications to PROSTINE® (vaginal gel of dinoprostone, cervical ripening agent)
* Contra-indications for using oxytocin
* Woman in labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1494 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Cesarean delivery rate | Up to 2 days after intervention
  The main outcome is the rate of caesarean delivery, whatever the indication of the caesarean delivery

SECONDARY OUTCOMES:
Time from intervention to delivery in hours | Up to 2 days after intervention
The proportion of women who delivered within 12 hours of the intervention | Up to 12 hours after intervention
Maternal satisfaction, assessed with the self administered ACE Questionnaire for Assessing Childbirth Experience (QACE) | 1 month
The proportion of women who require induction with oxytocin (for women in the control group) | Up to 2 days after intervention
The indications of caesarean in case of caesarean delivery | Up to 2 days after intervention
The proportion of women with an instrumental delivery | Up to 2 days after intervention
The indications for the use of instruments in case of instrumental delivery | Up to 2 days after intervention
The proportion of women suspected of per-partum infection | Up to 2 days after intervention
The proportion of women with post-partum haemorrhage | Up to 1 day after delivery
The proportion of women with severe Post-partum haemorrhage | Up to 2 days after intervention
The proportion of women with anal sphincter injury at delivery | Up to 2 days after intervention
The proportion of women who need blood transfusion | Up to 2 days after intervention
The proportion of women who need for antibiotics | Up to 2 days after intervention
The proportion of women admitted to intensive care unit | Up to 2 days after intervention

OTHER OUTCOMES:
Number and rate of children with an Apgar score under 7 | Up to 2 days after intervention
Number and rate of children with neonatal acidosis defined as umbilical arterial pH <7,00 | Up to 2 days after intervention
Number and rate of children with early neonatal infection | Up to 7 days after delivery
Number and rate of children admitted in an intensive care unit | Up to 7 days after delivery
Proportion of incremental cost-effect pairs | Up to 8 weeks
  Health economic outcome

CONTACTS AND LOCATIONS:
Overall Officials: Caroline DIGUISTO, MD, Study Director
Locations (12):
- France (12):
  - Gynaecology-obstetrics, University Hospital, Angers, Angers
  - Gynaecology-obstetrics, University Hospital, Bordeaux, Bordeaux
  - Gynaecology-obstetrics, University Hospital, Brest, Brest
  - Gynaecology-obstetrics, University Hospital, Clermont-Ferrand, Clermont-Ferrand
  - Gynaecology-obstetrics, Hospital St Joseph, Marseille, Marseille
  - Gynaecology-obstetrics, University Hospital, Nancy, Nancy
  - Gynaecology-obstetrics, University Hospital, Nantes, Nantes
  - Gynaecology-obstetrics, University Hospital, Orléans, Orléans
  - Gynaecology-obstetrics, Port Royal Maternity Hospital, Paris, Paris
  - Gynaecology-obstetrics, University Hospital, Poitiers, Poitiers
  - Gynaecology-obstetrics, University Hospital, Saint Etienne, Saint-Etienne
  - Gynaecology-obstetrics, University Hospital, Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data after de-identification can be obtained by contacting the corresponding author
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available immediately following publication and ending in 5 years
Access Criteria: Contact with the corresponding author

REFERENCES:
- [Derived] De Berti M, Le Gouge A, Monmousseau F, Gallot D, Sentilhes L, Winer N, Legendre G, Desbriere R, Girault A, Pozzi J, Gachon B, Barjat T, Perrotin F, Brunet-Houdard S, Diguisto C; Groupe de Recherche en Gynecologie Obstetrique. Oxytocin versus prostaglandins for labour Induction of women with an unfavourable cervix after 24 hours of cervical ripening (OPIC): protocol for an open multicentre randomised non-inferiority trial. BMJ Open. 2023 Apr 17;13(4):e058282. doi: 10.1136/bmjopen-2021-058282. PMID 37068892